CLINICAL TRIAL: NCT01690065
Title: Nilotinib Combined by Chemotherapy for Myeloid Blastic Phase of Chronic Myeloid Leukemia or Bcr-abl Positive Acute Myeloid Leukemia
Brief Title: Nilotinib-Chemotherapy in CML Myeloid BP or Bcr-abl(+) AML
Acronym: NICE-BORA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulsan University Hospital (Other)
Collaborators: The Korean Society of Hematology CML working party (Unknown)
Responsible Party: Principal Investigator, Hawk Kim, Associate Professor, Ulsan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AKR07T
Record Dates: First submitted 2012-09-11; First posted 2012-09-21 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Myeloid Leukemia in Myeloid Blast Crisis; Untreated Adult Acute Myeloid Leukemia
Keywords: chronic myeloid leukemia; myeloid blastic phase; bcr-abl(+) acute myeloid leukemia; nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib+AD induction (Experimental): Nilotinib plus AD induction chemotherapy
  * AD regimen : Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 7 days (D 1-7) plus Daunorubicin 90 mg/m2/day iv daily for 3 days (D 1-3)
  * Nilotinib 400mg bid PO (continuous without interruption from D8 of induction chemotherapy)
  * Re-induction chemotherapy AD regimen : Cytarabine 200 mg/m2/day by continuous iv infusion over 24 hours daily for 5 days (D 1-5) plus Daunorubicin 45 mg/m2/day iv daily for 2 days (D 1-2)
  Interventions: Drug: Nilotinib+AD induction

INTERVENTIONS:
Drug: Nilotinib+AD induction — • Post-remission consolidation chemotherapy
  * 4 courses of high-dose cytarabine will be given as post-remission therapy. Cytarabine 3 g/m2 will be administered in a 3-hour iv infusion every 12 hours on days 1, 3, and 5 (a total of six doses per course).
  * Nilotinib 400mg bid PO will be administered continuously during consolidation chemotherapy and for 2 years after the consolidation therapy or until allogeneic hematopoietic stem cell transplantation
  Other Names: Tasigna

SUMMARY:
The current standard therapy in previously untreated adults with chronic phase (CP) of CML is imatinib and the result of long-term follow-up of IRIS study proves that imatinib for CML CP is reasonable therapy.(1, 2) However, some patients were initially diagnosed as advanced CML, accelerated phase (AP) or blastic phase (BP). Various chemotherapies were tried and were found that there were no highly effective chemotherapies for CML BP.(3-11) Imatinib in patients with these advanced CML is also disappointing because of low response rates as well as short response duration, and sudden transformation to BC is found even in initial CML CP patients. (12-17). Recent studies showed that nilotinib or dasatinib is better than imatinib in terms of rapid response and higher molecular response in newly diagnosed CML patients.(18-21) More potent bcr-abl suppression of nilotinib is supposed to be more active than imatinib even in patients with advanced CML. However, nilotinib in patients with imatinib-resistant or -intolerant CML BP showed low hematologic response and major cytogenetic response.(22, 23)

DETAILED DESCRIPTION:
1. IMATINIB COMBINED WITH CHEMOTHERAPY FOR PHYLADELPHIA POSITIVE ACUTE LYMPHOBLASTIC LYMPHOMA (PH+ ALL) The trials combining imatinib with high-dose chemotherapy were successfully resulting in high response rate and longer survival and a role for bridging therapy to allogeneic hematopoietic stem cell transplantation (alloHSCT) by means of concurrent or alternating regimen in patients with Philadelphia-positive (Ph+) acute lymphoblastic leukemia (ALL).(24-29) Current combination therapy of imatinib and chemotherapy became standard therapy of Ph+ ALL and new 2nd generation TKIs are investigating. These experiences may be translated into the treatment of CML BP.
2. HIGH-DOSE DAUNORUBICIN IN ACUTE MYELOID LEUKEMIA (AML) INDUCTION CHEMOTHERAPY Two recently published papers of randomized trials comparing standard dose daunorubicin (45 mg/m2 for 3 days) and high dose daunorubicin (90 mg/m2 for 3 days) demonstrated improved CR rate and survival with high dose daunorubicin in younger (60 years or younger) and older (over 60 years) patients, respectively.(30, 31) Therefore high-dose daunorubicin can be applied safely and effectively to the treatment of CML BP.
3. NILOTINIB COMBINED WITH CHEMOTHERAPY FOR PHYLADELPHIA POSITIVE CML MYELOID BLASTIC PHASE (MBP) OR PHYLADELPHIA POSITIVE AML We will try 2nd generation TKI, nilotinib and high-dose daunorubicin induction chemotherapy combination to find out the combination therapy can improve response rate and survival in patients with CML MBP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously-untreated patients having bcr-abl gene rearrangement (or t(9;22)) and 20% or more of myeloid blasts in bone marrow and/or blood, or converted CML CP/AP to MBP after initial imatinib treatment.
* 15 years old or older, but 65 years or younger
* Adequate performance status (Karnofsky score of 50 or more)
* Adequate hepatic and renal function (AST, ALT, bilirubin and creatinine < 2.5 x upper normal limit). Elevation of AST or ALT due to hepatic infiltration of leukemic cells will be permitted.
* Adequate cardiac function (left ventricular ejection fraction of 45% or more on heart scan or echocardiogram)
* Signed and dated informed consent must be obtained.

Exclusion Criteria:

* Patients without bcr-abl gene rearrangement
* Acute lymphoblastic leukemia with bcr-abl gene rearrangement or t(9;22)
* Any previous history of TKIs except for imatinib in CML CP.
* Therapy-related leukemia or leukemia after myelodysplastic syndrome.
* Patients with CNS leukemia
* Patients with primary granulocytic sarcoma without bone marrow involvement
* Prior chemotherapy for leukemia or anthracycline treatment for any malignancy. Hydroxyurea for reduction of leukemic cell burden before induction chemotherapy will be permitted.
* Presence of significant active infection
* Presence of uncontrolled bleeding
* Significant cardiovascular disease including myocardial infarction within previous 6 months
* Cardiac dysfunction: LVEF < 45% or institutional lower normal range (any higher value of them) by echocardiogram or MUGA scan; Long QT syndrome or its family history; Clinically significant resting bradycardia (<50 beats/minute); QTc > 450 msec (by QTcF formula) on baseline ECG . If QTcF > 450 msec and electrolytes are abnormal, retest QTc after the correction of electrolytes; Myocardial infarction within 12 months; Other clinically significant cardiac diseases (for example, unstable angina, congestive heart failure, uncontrolled hypertension or uncontrolled arrhythmia)
* Chronic or acute hepatic disease, pancreatic disease or severe renal disease
* Severe or life-threatening other medical conditions
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible History of congenital or acquired coagulopathy unrelated to malignancy
* Pregnancy issues: (a) pregnant woman, (b) lactating woman, (c) reproductive woman who does not confirm negative baseline pregnancy test (d) man or reproductive woman who cannot continue an appropriate contraceptive method (postmenopausal woman who has no menstruation for last 12 months is considered as non-reproductive)
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)
* History of non-compliance or patient who cannot sign informed consent
* Hypersensitivity to nilotinib or any of the experience
* Concurrent medications (Gastrointestinal dysfunction that can significantly change the absorption of test drug; - Strong CYP3A4 inhibitor and cannot stop or change the medication before starting study; Medication to prolong QT interval and cannot stop or change the medication before starting study) • The capsules contain lactose, and nilotinib is therefore not recommended for patients with rare hereditary problems of galactose intolerance, severe lactase deficiency or glucose-galactose malabsorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2012-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | Within 8 weeks after induction therapy
  Primary purpose of this study is to define the efficacy of combined chemotherapy and nilotinib in chronic myeloid leukemia (CML) myeloid blastic phase (MBP) and bcr-abl positive acute myeloid leukemia (AML). The efficacy will be evaluated by complete remission (CR) rate.

SECONDARY OUTCOMES:
Safety | Within 8 weeks after induction therapy
  * This study will also evaluate the safety of nilotinib and chemotherapy combination therapy.
  * CTCAE ver. 4.03 will be used for safety measurement.
Time-dependent variables | at least 2 years
  • This study will evaluate the impacts of nilotinib combined with chemotherapy on duration of CR, relapse-free survival (RFS), event-free survival (EFS), and overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Hawk Kim, M.D., Ph.D., Principal Investigator — Ulsan University Hospital, University of Ulsan College of Medicine
Locations (2):
- South Korea (2):
  - Seoul St Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Background] O'Brien SG, Guilhot F, Larson RA, Gathmann I, Baccarani M, Cervantes F, Cornelissen JJ, Fischer T, Hochhaus A, Hughes T, Lechner K, Nielsen JL, Rousselot P, Reiffers J, Saglio G, Shepherd J, Simonsson B, Gratwohl A, Goldman JM, Kantarjian H, Taylor K, Verhoef G, Bolton AE, Capdeville R, Druker BJ; IRIS Investigators. Imatinib compared with interferon and low-dose cytarabine for newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2003 Mar 13;348(11):994-1004. doi: 10.1056/NEJMoa022457. PMID 12637609
- [Background] Hochhaus A, O'Brien SG, Guilhot F, Druker BJ, Branford S, Foroni L, Goldman JM, Muller MC, Radich JP, Rudoltz M, Mone M, Gathmann I, Hughes TP, Larson RA; IRIS Investigators. Six-year follow-up of patients receiving imatinib for the first-line treatment of chronic myeloid leukemia. Leukemia. 2009 Jun;23(6):1054-61. doi: 10.1038/leu.2009.38. Epub 2009 Mar 12. PMID 19282833
- [Background] Bauduer F, Delmer A, Blanc MC, Delmas-Marsalet B, Cadiou M, Rio B, Marie JP, Zittoun R. Treatment of chronic myelogenous leukemia in blast crisis and in accelerated phase with high- or intermediate-dose cytosine arabinoside and amsacrine. Leuk Lymphoma. 1993 Jun;10(3):195-200. doi: 10.3109/10428199309145883. PMID 8220118
- [Background] Coleman M, Silver RT, Pajak TF, Cavalli F, Rai KR, Kostinas JE, Glidewell O, Holland JF. Combination chemotherapy for terminal-phase chronic granulocytic leukemia: cancer and leukemia group B studies. Blood. 1980 Jan;55(1):29-36. PMID 6927956
- [Background] Dutcher JP, Eudey L, Wiernik PH, Paietta E, Bennett JM, Arlin Z, Kellermeyer R, Rowe J, O'Connell M, Oken M, et al. Phase II study of mitoxantrone and 5-azacytidine for accelerated and blast crisis of chronic myelogenous leukemia: a study of the Eastern Cooperative Oncology Group. Leukemia. 1992 Aug;6(8):770-5. PMID 1379312
- [Background] Dutcher JP, Lee S, Paietta E, Bennett JM, Stewart JA, Wiernik PH. Phase II study of carboplatin in blast crisis of chronic myeloid leukemia: Eastern Cooperative Oncology Group Study E1992. Leukemia. 1998 Jul;12(7):1037-40. doi: 10.1038/sj.leu.2401056. PMID 9665187
- [Background] Feldman EJ, Alberts DS, Arlin Z, Ahmed T, Mittelman A, Baskind P, Peng YM, Baier M, Plezia P. Phase I clinical and pharmacokinetic evaluation of high-dose mitoxantrone in combination with cytarabine in patients with acute leukemia. J Clin Oncol. 1993 Oct;11(10):2002-9. doi: 10.1200/JCO.1993.11.10.2002. PMID 8410125
- [Background] Giles FJ, Feldman EJ, Roboz GJ, Larson RA, Mamus SW, Cortes JE, Verstovsek S, Faderl S, Talpaz M, Beran M, Albitar M, O'Brien SM, Kantarjian HM. Phase II study of troxacitabine, a novel dioxolane nucleoside analog, in patients with untreated or imatinib mesylate-resistant chronic myelogenous leukemia in blastic phase. Leuk Res. 2003 Dec;27(12):1091-6. doi: 10.1016/s0145-2126(03)00094-8. PMID 12921945
- [Background] Kantarjian HM, O'Brien S, Cortes J, Giles FJ, Faderl S, Issa JP, Garcia-Manero G, Rios MB, Shan J, Andreeff M, Keating M, Talpaz M. Results of decitabine (5-aza-2'deoxycytidine) therapy in 130 patients with chronic myelogenous leukemia. Cancer. 2003 Aug 1;98(3):522-8. doi: 10.1002/cncr.11543. PMID 12879469
- [Background] Koller CA, Miller DM. Preliminary observations on the therapy of the myeloid blast phase of chronic granulocytic leukemia with plicamycin and hydroxyurea. N Engl J Med. 1986 Dec 4;315(23):1433-8. doi: 10.1056/NEJM198612043152301. PMID 2431313
- [Background] O'Brien S, Kantarjian H, Keating M, Beran M, Koller C, Robertson LE, Hester J, Rios MB, Andreeff M, Talpaz M. Homoharringtonine therapy induces responses in patients with chronic myelogenous leukemia in late chronic phase. Blood. 1995 Nov 1;86(9):3322-6. PMID 7579434
- [Background] Jabbour E, Kantarjian H, O'Brien S, Rios MB, Abruzzo L, Verstovsek S, Garcia-Manero G, Cortes J. Sudden blastic transformation in patients with chronic myeloid leukemia treated with imatinib mesylate. Blood. 2006 Jan 15;107(2):480-2. doi: 10.1182/blood-2005-05-1816. Epub 2005 Sep 29. PMID 16195326
- [Background] Kantarjian HM, Cortes J, O'Brien S, Giles FJ, Albitar M, Rios MB, Shan J, Faderl S, Garcia-Manero G, Thomas DA, Resta D, Talpaz M. Imatinib mesylate (STI571) therapy for Philadelphia chromosome-positive chronic myelogenous leukemia in blast phase. Blood. 2002 May 15;99(10):3547-53. doi: 10.1182/blood.v99.10.3547. PMID 11986206
- [Background] Morimoto A, Ogami A, Chiyonobu T, Takanashi M, Sugimoto T, Imamura T, Ishida H, Yoshihara T, Imashuku S. Early blastic transformation following complete cytogenetic response in a pediatric chronic myeloid leukemia patient treated with imatinib mesylate. J Pediatr Hematol Oncol. 2004 May;26(5):320-2. doi: 10.1097/00043426-200405000-00013. PMID 15111787
- [Background] Pavlu J, Czepulkowski B, Kaczmarski R, Jan-Mohamed R. Early blastic transformation with CNS infiltration in a patient with chronic myeloid leukaemia treated with imatinib. Lancet Oncol. 2005 Feb;6(2):128. doi: 10.1016/S1470-2045(05)01744-4. No abstract available. PMID 15683824
- [Background] Sureda A, Carrasco M, de Miguel M, Martinez JA, Conde E, Sanz MA, Diaz-Mediavilla J, Sierra J. Imatinib mesylate as treatment for blastic transformation of Philadelphia chromosome positive chronic myelogenous leukemia. Haematologica. 2003 Nov;88(11):1213-20. PMID 14607749
- [Background] Palandri F, Castagnetti F, Alimena G, Testoni N, Breccia M, Luatti S, Rege-Cambrin G, Stagno F, Specchia G, Martino B, Levato L, Merante S, Liberati AM, Pane F, Saglio G, Alberti D, Martinelli G, Baccarani M, Rosti G. The long-term durability of cytogenetic responses in patients with accelerated phase chronic myeloid leukemia treated with imatinib 600 mg: the GIMEMA CML Working Party experience after a 7-year follow-up. Haematologica. 2009 Feb;94(2):205-12. doi: 10.3324/haematol.13529. Epub 2009 Jan 14. PMID 19144656
- [Background] Saglio G, Kim DW, Issaragrisil S, le Coutre P, Etienne G, Lobo C, Pasquini R, Clark RE, Hochhaus A, Hughes TP, Gallagher N, Hoenekopp A, Dong M, Haque A, Larson RA, Kantarjian HM; ENESTnd Investigators. Nilotinib versus imatinib for newly diagnosed chronic myeloid leukemia. N Engl J Med. 2010 Jun 17;362(24):2251-9. doi: 10.1056/NEJMoa0912614. Epub 2010 Jun 5. PMID 20525993
- [Background] Kantarjian H, Shah NP, Hochhaus A, Cortes J, Shah S, Ayala M, Moiraghi B, Shen Z, Mayer J, Pasquini R, Nakamae H, Huguet F, Boque C, Chuah C, Bleickardt E, Bradley-Garelik MB, Zhu C, Szatrowski T, Shapiro D, Baccarani M. Dasatinib versus imatinib in newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2010 Jun 17;362(24):2260-70. doi: 10.1056/NEJMoa1002315. Epub 2010 Jun 5. PMID 20525995
- [Background] Cortes JE, Jones D, O'Brien S, Jabbour E, Konopleva M, Ferrajoli A, Kadia T, Borthakur G, Stigliano D, Shan J, Kantarjian H. Nilotinib as front-line treatment for patients with chronic myeloid leukemia in early chronic phase. J Clin Oncol. 2010 Jan 20;28(3):392-7. doi: 10.1200/JCO.2009.25.4896. Epub 2009 Dec 14. PMID 20008621
- [Background] Rosti G, Palandri F, Castagnetti F, Breccia M, Levato L, Gugliotta G, Capucci A, Cedrone M, Fava C, Intermesoli T, Cambrin GR, Stagno F, Tiribelli M, Amabile M, Luatti S, Poerio A, Soverini S, Testoni N, Martinelli G, Alimena G, Pane F, Saglio G, Baccarani M; GIMEMA CML Working Party. Nilotinib for the frontline treatment of Ph(+) chronic myeloid leukemia. Blood. 2009 Dec 3;114(24):4933-8. doi: 10.1182/blood-2009-07-232595. Epub 2009 Oct 12. PMID 19822896
- [Background] Fava C, Kantarjian HM, Jabbour E, O'Brien S, Jain N, Rios MB, Garcia-Manero G, Ravandi F, Verstovsek S, Borthakur G, Shan J, Cortes J. Failure to achieve a complete hematologic response at the time of a major cytogenetic response with second-generation tyrosine kinase inhibitors is associated with a poor prognosis among patients with chronic myeloid leukemia in accelerated or blast phase. Blood. 2009 May 21;113(21):5058-63. doi: 10.1182/blood-2008-10-184960. Epub 2009 Mar 12. PMID 19282457
- [Background] Jabbour E, Cortes J, Kantarjian H. Nilotinib for the treatment of chronic myeloid leukemia: An evidence-based review. Core Evid. 2010 Jun 15;4:207-13. doi: 10.2147/ce.s6003. PMID 20694077
- [Background] Lee KH, Lee JH, Choi SJ, Lee JH, Seol M, Lee YS, Kim WK, Lee JS, Seo EJ, Jang S, Park CJ, Chi HS. Clinical effect of imatinib added to intensive combination chemotherapy for newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia. Leukemia. 2005 Sep;19(9):1509-16. doi: 10.1038/sj.leu.2403886. PMID 16034462
- [Background] Lee S, Kim YJ, Min CK, Kim HJ, Eom KS, Kim DW, Lee JW, Min WS, Kim CC. The effect of first-line imatinib interim therapy on the outcome of allogeneic stem cell transplantation in adults with newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood. 2005 May 1;105(9):3449-57. doi: 10.1182/blood-2004-09-3785. Epub 2005 Jan 18. PMID 15657178
- [Background] Potenza L, Luppi M, Riva G, Marasca R, Martinelli S, Torelli G. Efficacy of imatinib mesylate as maintenance therapy in adults with acute lymphoblastic leukemia in first complete remission. Haematologica. 2005 Sep;90(9):1275-7. PMID 16154854
- [Background] Rea D, Legros L, Raffoux E, Thomas X, Turlure P, Maury S, Dupriez B, Pigneux A, Choufi B, Reman O, Stephane D, Royer B, Vigier M, Ojeda-Uribe M, Recher C, Dombret H, Huguet F, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chronique; Group for Research in Adult Acute Lymphoblastic Leukemia. High-dose imatinib mesylate combined with vincristine and dexamethasone (DIV regimen) as induction therapy in patients with resistant Philadelphia-positive acute lymphoblastic leukemia and lymphoid blast crisis of chronic myeloid leukemia. Leukemia. 2006 Mar;20(3):400-3. doi: 10.1038/sj.leu.2404115. PMID 16437142
- [Background] Thomas DA, Faderl S, Cortes J, O'Brien S, Giles FJ, Kornblau SM, Garcia-Manero G, Keating MJ, Andreeff M, Jeha S, Beran M, Verstovsek S, Pierce S, Letvak L, Salvado A, Champlin R, Talpaz M, Kantarjian H. Treatment of Philadelphia chromosome-positive acute lymphocytic leukemia with hyper-CVAD and imatinib mesylate. Blood. 2004 Jun 15;103(12):4396-407. doi: 10.1182/blood-2003-08-2958. Epub 2003 Oct 9. PMID 14551133
- [Background] Wassmann B, Pfeifer H, Goekbuget N, Beelen DW, Beck J, Stelljes M, Bornhauser M, Reichle A, Perz J, Haas R, Ganser A, Schmid M, Kanz L, Lenz G, Kaufmann M, Binckebanck A, Bruck P, Reutzel R, Gschaidmeier H, Schwartz S, Hoelzer D, Ottmann OG. Alternating versus concurrent schedules of imatinib and chemotherapy as front-line therapy for Philadelphia-positive acute lymphoblastic leukemia (Ph+ ALL). Blood. 2006 Sep 1;108(5):1469-77. doi: 10.1182/blood-2005-11-4386. Epub 2006 Apr 25. PMID 16638934
- [Background] Fernandez HF, Sun Z, Yao X, Litzow MR, Luger SM, Paietta EM, Racevskis J, Dewald GW, Ketterling RP, Bennett JM, Rowe JM, Lazarus HM, Tallman MS. Anthracycline dose intensification in acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1249-59. doi: 10.1056/NEJMoa0904544. PMID 19776406
- [Background] Lowenberg B, Ossenkoppele GJ, van Putten W, Schouten HC, Graux C, Ferrant A, Sonneveld P, Maertens J, Jongen-Lavrencic M, von Lilienfeld-Toal M, Biemond BJ, Vellenga E, van Marwijk Kooy M, Verdonck LF, Beck J, Dohner H, Gratwohl A, Pabst T, Verhoef G; Dutch-Belgian Cooperative Trial Group for Hemato-Oncology (HOVON); German AML Study Group (AMLSG); Swiss Group for Clinical Cancer Research (SAKK) Collaborative Group. High-dose daunorubicin in older patients with acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1235-48. doi: 10.1056/NEJMoa0901409. PMID 19776405
- [Background] Wassmann B, Pfeifer H, Stadler M, Bornhauser M, Bug G, Scheuring UJ, Bruck P, Stelljes M, Schwerdtfeger R, Basara N, Perz J, Bunjes D, Ledderose G, Mahlberg R, Binckebanck A, Gschaidmeier H, Hoelzer D, Ottmann OG. Early molecular response to posttransplantation imatinib determines outcome in MRD+ Philadelphia-positive acute lymphoblastic leukemia (Ph+ ALL). Blood. 2005 Jul 15;106(2):458-63. doi: 10.1182/blood-2004-05-1746. Epub 2005 Apr 7. PMID 15817679